CLINICAL TRIAL: NCT02825043
Title: Effect of High-Flow Nasal Cannula (HFNC) on the Breathlessness, Cough, and Sputum Scale (BCSS), in Patients With Stable Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: HFNC Effect on BCSS in Patients With COPD
Acronym: COPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment and unable to meet enrollment targets
Sponsor: University of Oklahoma (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6410
Record Dates: First submitted 2016-06-29; First posted 2016-07-07 (Estimated); Results first posted 2020-06-29 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High Flow Nasal Cannula Participants (Experimental): High Flow Nasal Cannula Participants will be their own control, they will be in study for 3 months prior to receiving equipment and then will be studied for 3 additional months on study.
  Interventions: Device: High-Flow Nasal Cannula

INTERVENTIONS:
Device: High-Flow Nasal Cannula — This is a humidified oxygen delivery system.
  Other Names: AIRVO 2 Series Humidifier

SUMMARY:
The primary objective of this study is to look for a correlation between the use of high-flow nasal cannula in the outpatient setting in patients with previous chronic obstructive pulmonary disease exacerbation and the change in their Breathlessness, Cough, and Sputum Scale score. The hypothesis is that home use of high-flow nasal cannula will lead to a reduction in Breathlessness, Cough, and Sputum Scale score by 1.3.

DETAILED DESCRIPTION:
This is a prospective pilot study. Targeted population include patients with chronic obstructive pulmonary disease , non-oxygen dependent, with a baseline normal bicarbonate on previous lab (within 6 months of enrollment). Patients will be randomly selected to be part of the study sample. Recruitment will occur in both inpatient and outpatient settings. An email briefly explaining the objectives of the study will be sent to Internal Medicine residents and Pulmonary Critical Care fellows to help in patients' recruitment. Patients will be enrolled in the study only after being seen by Dr. Abdo or Dr. Allen. The study is expected to finish by the end of January 2017 or twelve months post institutional review board approval. Patients will be recruited and enrolled over six months, and the collected data will be analyzed six months after the last patient was included in the study. The study will target a study sample of 30 as detailed in the statistical analysis section, where patients will be their own control (3 months without high-flow nasal cannula followed by 3 months with high-flow nasal cannula).

ELIGIBILITY:
Inclusion Criteria:

One previous chronic obstructive pulmonary disease exacerbation in last year.

Exclusion Criteria:

Can not be oxygen dependant PaCO2 < 60

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Allen, MD, Principal Investigator — OUMC
Locations (1):
- University of Oklahoma, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
Will share data as a cohort for other investigators, but will not share individual participant data.

REFERENCES:
- [Background] Spoletini G, Alotaibi M, Blasi F, Hill NS. Heated Humidified High-Flow Nasal Oxygen in Adults: Mechanisms of Action and Clinical Implications. Chest. 2015 Jul;148(1):253-261. doi: 10.1378/chest.14-2871. PMID 25742321
- [Background] Nishimura M. High-flow nasal cannula oxygen therapy in adults. J Intensive Care. 2015 Mar 31;3(1):15. doi: 10.1186/s40560-015-0084-5. eCollection 2015. PMID 25866645
- [Background] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Background] Braunlich J, Seyfarth HJ, Wirtz H. Nasal High-flow versus non-invasive ventilation in stable hypercapnic COPD: a preliminary report. Multidiscip Respir Med. 2015 Sep 3;10(1):27. doi: 10.1186/s40248-015-0019-y. eCollection 2015. PMID 26339486
- [Background] Braunlich J, Beyer D, Mai D, Hammerschmidt S, Seyfarth HJ, Wirtz H. Effects of nasal high flow on ventilation in volunteers, COPD and idiopathic pulmonary fibrosis patients. Respiration. 2013;85(4):319-25. doi: 10.1159/000342027. Epub 2012 Nov 1. PMID 23128844
- [Background] Nilius G, Franke KJ, Domanski U, Ruhle KH, Kirkness JP, Schneider H. Effects of nasal insufflation on arterial gas exchange and breathing pattern in patients with chronic obstructive pulmonary disease and hypercapnic respiratory failure. Adv Exp Med Biol. 2013;755:27-34. doi: 10.1007/978-94-007-4546-9_4. PMID 22826046
- [Background] Leidy NK, Rennard SI, Schmier J, Jones MK, Goldman M. The breathlessness, cough, and sputum scale: the development of empirically based guidelines for interpretation. Chest. 2003 Dec;124(6):2182-91. doi: 10.1378/chest.124.6.2182. PMID 14665499

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Flow Nasal Cannula Participants
Started | 6
Completed | 2
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | High Flow Nasal Cannula Participants
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex Not Collected | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Changes in Breathlessness, Cough and Sputum Scale (BCSS)
Description: The Changes in Breathlessness, Cough and Sputum Scale (BCSS) is a three question measure consisting of three questions, each rated on a scale of "0" to "4", with a total possible score ranging from 0-12. Zero equals no difficulty and four equals severe difficulty or constant problem. A lower score on the scale is a better outcome.
Time Frame: 6 months
Population: Four (4) participants were lost to follow-up and no data was collected. Two (2) participants returned BCSS scores at which time, baseline data was not collected due to decision to terminate study. Baseline data is required to calculate change in BCSS.
Arm/Group | High Flow Nasal Cannula Participants
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in Number of Chronic Obstructive Pulmonary Disease Exacerbations Per Month
Description: The number of chronic obstructive pulmonary disease exacerbations per month will be monitored throughout the study. A lower number of chronic obstructive pulmonary disease exacerbations are considered improvement.
Time Frame: 6 months
Population: Four (4) participants were lost to follow-up and no data was collected on those participants. Data was not collected on remaining two (2) participants for this outcome measure.
Arm/Group | High Flow Nasal Cannula Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | High Flow Nasal Cannula Participants
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 1/5
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Flow Nasal Cannula Participants (N=5)
Condensation in tubing (Product Issues) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-29): https://cdn.clinicaltrials.gov/large-docs/43/NCT02825043/Prot_SAP_000.pdf